CLINICAL TRIAL: NCT01474889
Title: Effect of Real-Time Continuous Glucose Monitoring on Glucose Counterregulation in Long Standing Type 1 Diabetes
Brief Title: Glucose Counterregulation in Long Standing Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael R. Rickels, MD, MS, Professor of Medicine, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 814114; R01DK091331-01 (NIH)
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Hypoglycemia Unawareness; Type 1 Diabetes; Healthy
Keywords: Hypoglycemia, Unawareness, RT-CGM, Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Unconsciousness

STUDY DESIGN:
Intervention Model Description: Hypoglycemia Unaware T1 Diabetics & 2 Control Groups. Non-Diabetics & T1Ds With Intact Awareness.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypoglycemia Unaware T1 Diabetes RT-CGM (Experimental): This arm is the intervention group. It consists of participants with type 1 diabetes complicated by hypoglycemia unawareness. Patients wore an RT-CGM for 18 months. We studied glucose production and symptom generation during insulin-induced hypoglycemia (metabolic testing) by subjecting this intervention group to a pair of metabolic clamps (hypoglycemic and euglycemic) at baseline, at 6 months and at 18 months to determine if hypoglycemia avoidance can reverse unawareness.
  Please note: Arms are not assigned to the two control groups (non-diabetics and T1Ds with intact awareness) in ct.gov as they are only used as a baseline for clinical significance. Neither group wore a CGM nor are they analyzed at 6-month and 18-month time-points.
  Interventions: Device: RT-CGM

INTERVENTIONS:
Device: RT-CGM — Each device is approximately the size of a pager and transmits with a subcutaneously placed sensor consisting of a 21 - 26 gauge needle 5 - 12 mm in length. Sensors are placed using sterile precautions and changed every 3 - 7 days depending on the manufacturers' instructions. All devices are approved as adjunctive tools to blood glucose monitoring that will be continued at least 4 times daily, before each meal and at bedtime.
  Other Names: DexCom SEVEN PLUS, Guardian R-T, or FreeStyle Navigator.

SUMMARY:
Enrollment for this study is complete.

This study is designed to determine if use of a real-time continuous glucose monitor (RT-CGM) can reverse defective Glucose counter regulation and hypoglycemia unawareness in long standing type 1 diabetes.

DETAILED DESCRIPTION:
The present protocol is designed to determine whether strict hypoglycemia avoidance by real-time continuous glucose monitoring (RT-CGM), can restore endogenous glucose production in response to hypoglycemia in patients with long standing disease. Twelve subjects with long standing type 1 diabetes complicated by hypoglycemia unawareness underwent assessment of the endogenous glucose production response to insulin-induced hypoglycemia using paired hyperinsulinemic euglycemic and hypoglycemic clamps with stable glucose isotope infusions before and at 6 and 18 months following initiation of RT-CGM. The primary analysis will be change in the endogenous glucose production response from before to 6 months following initiation of RT-CGM, and a secondary analysis will consider the persistence of any change at 18 months. The clinical significance of any determined changes in the endogenous glucose production response to insulin-induced hypoglycemia will be determined by comparison to responses obtained using paired hyperinsulinemic euglycemic and hypoglycemic clamps on one occasion in a matched control group of 12 subjects with long-standing type 1 diabetes but no hypoglycemia unawareness (GROUP 2) and in a matched control group of 12 nondiabetic subjects (GROUP 3).

Arms are not assigned to these two control groups in ct.gov as they were only used as a baseline for clinical significance. Neither group wore a CGM nor are they analyzed at 6-month and 18-month time-points. This said, for control group clarification, inclusion and exclusion criteria for each group is included in ct.gov

Hypoglycemia is a major barrier to the achievement of adequate glycemic control for most patients with insulin-dependent diabetes. Type 1 diabetic patients with absolute insulin deficiency (C-peptide negative) are at greatest risk for experiencing severe hypoglycemic events because the near total destruction of insulin producing islet β-cells produces an associated defect in glucagon secretion from neighboring α-cells. Such patients then depend on the sympathoadrenal system as a final defense against hypoglycemia, but unfortunately, recurrent episodes of hypoglycemia blunt sympathoadrenal activation and produce a syndrome of hypoglycemia unawareness that is associated with a twenty-fold increased risk of life-threatening hypoglycemia. Without intact islet or sympathoadrenal (especially epinephrine) responses to hypoglycemia, these patients cannot increase endogenous (primarily hepatic) glucose production to prevent or correct low blood glucose.

ELIGIBILITY:
Key Inclusion Criteria for intervention GROUP 1 (Long-standing T1D complicated by hypoglycemia unawareness)

1. Male and female subjects aged 25 to 70 years
2. Able to provide written informed consent and to comply with the protocol procedures
3. Clinical history compatible with type 1 diabetes with disease onset < 40 years of age OR onset ≥ 40 years and documented islet autoimmunity
4. Insulin-dependent for > 10 years
5. Absent C-peptide (< 0.3 ng/mL).
6. Involvement in intensive diabetes management defined as self-monitoring of glucose values no less than a mean of three times each day averaged over each week and by the administration of three or more insulin injections each day or insulin pump therapy under the direction of an endocrinologist, diabetologist, or diabetes specialist with at least 3 clinical evaluations during the previous 12 months.)
7. Hypoglycemia unawareness manifested by a Clarke score of 4 or more AND at least one of the following:

   * HYPO score greater than or equal to the 90th percentile (1047); OR marked glycemic lability defined by a glycemic lability index (LI) score greater than or equal to the 90th percentile (433 mmol/l2/h·wk-1); OR
   * A composite of a HYPO score greater than or equal to the 75th percentile (423) and a LI greater than or equal to the 75th percentile (329).
8. At least one episode of severe hypoglycemia in the past 12 months defined as an event with symptoms or signs compatible with hypoglycemia in which the subject was unable to treat him/herself and which was associated with either a blood glucose level < 54 mg/dl [3.0 mmol/L] or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration; OR documented > 5% time spent in the hypoglycemic range (glucose < 60 mg/dl) by 72-hour blinded CGM.

Key Inclusion Criteria for control GROUP 2 (Long-standing T1D with intact hypoglycemia awareness)

1. Male and female subjects aged 25 to 70 years.
2. Able to provide written informed consent and to comply with the procedures of the study protocol.
3. Clinical history compatible with type 1 diabetes with disease onset < 40 years of age
4. Insulin-dependent for > 10 years
5. Absent C-peptide (< 0.3 ng/mL).
6. Involvement in intensive diabetes management defined as the use of basal-bolus insulin analog delivery by multi-dose injection (MDI) or continuous subcutaneous insulin infusion (CSII) together with self-monitoring of blood glucose values four or more times daily, without continuous glucose monitoring (CGM), under the direction of an endocrinologist, diabetologist, or diabetes nurse practitioner with at least 3 clinical evaluations during the previous 12 months.
7. Intact hypoglycemia awareness indicated by a Clarke score of 3 or less.
8. No episodes of severe hypoglycemia in the past 3 years.

Key Inclusion Criteria for control GROUP 3 (Non-diabetic controls)

1. Male and female subjects aged 25 to 70 years.
2. Subjects who are able to provide written informed consent and to comply with the procedures of the study protocol.
3. No history of diabetes.

Key Exclusion Criteria for ALL 3 groups

1. Body mass index (BMI) greater than 38 kg/m2.
2. Insulin requirement of more than 1.0 IU/kg/day.
3. HbA1c greater than 10%.
4. Untreated proliferative diabetic retinopathy.
5. SBP greater than 160 mmHg or DBP greater than 100 mmHg.
6. Glomerular filtration rate (GFR) less than 55 ml/min/1.73 m-squared
7. Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study.
8. Baseline hemoglobin less than 11 g/dl in women and less than12 g/dl in men.
9. Severe co-existing cardiac disease
10. Persistent elevation of liver function tests greater than 1.5 upper normal limits
11. Hyperlipidemia despite medical therapy
12. Receiving treatment for a medical condition requiring chronic use of systemic steroids
13. Presence of a seizure disorder not attributable to hypoglycemia.
14. Untreated hypothyroidism, Addisons disease, or Celiac disease.
15. Treatment with any anti-diabetic medication other than insulin within 4 weeks of enrollment.
16. Use of RT-CGM (continuous glucose monitor) within last 4 weeks.

    * Non-diabetic patients do not need to meet any of the glucose criteria.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-10; Primary Completion 2016-05 (Actual); Study Completion 2021-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Rickels, M.D., M.S., Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Clinical and Translational Research Center, Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Rodebaugh Diabetes Center, University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania - Institute for Diabetes, Obesity and Metabolism, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hypoglycemia in the Diabetes Control and Complications Trial. The Diabetes Control and Complications Trial Research Group. Diabetes. 1997 Feb;46(2):271-86. PMID 9000705
- [Background] Cryer PE. Mechanisms of hypoglycemia-associated autonomic failure and its component syndromes in diabetes. Diabetes. 2005 Dec;54(12):3592-601. doi: 10.2337/diabetes.54.12.3592. PMID 16306382
- [Background] Pedersen-Bjergaard U, Pramming S, Heller SR, Wallace TM, Rasmussen AK, Jorgensen HV, Matthews DR, Hougaard P, Thorsteinsson B. Severe hypoglycaemia in 1076 adult patients with type 1 diabetes: influence of risk markers and selection. Diabetes Metab Res Rev. 2004 Nov-Dec;20(6):479-86. doi: 10.1002/dmrr.482. PMID 15386817
- [Background] Tanenberg R, Bode B, Lane W, Levetan C, Mestman J, Harmel AP, Tobian J, Gross T, Mastrototaro J. Use of the Continuous Glucose Monitoring System to guide therapy in patients with insulin-treated diabetes: a randomized controlled trial. Mayo Clin Proc. 2004 Dec;79(12):1521-6. doi: 10.4065/79.12.1521. PMID 15595336
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Tamborlane WV, Beck RW, Bode BW, Buckingham B, Chase HP, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Hirsch IB, Huang ES, Kollman C, Kowalski AJ, Laffel L, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer S, Wilson DM, Wolpert H, Wysocki T, Xing D. Continuous glucose monitoring and intensive treatment of type 1 diabetes. N Engl J Med. 2008 Oct 2;359(14):1464-76. doi: 10.1056/NEJMoa0805017. Epub 2008 Sep 8. PMID 18779236
- [Background] Hirsch IB, Abelseth J, Bode BW, Fischer JS, Kaufman FR, Mastrototaro J, Parkin CG, Wolpert HA, Buckingham BA. Sensor-augmented insulin pump therapy: results of the first randomized treat-to-target study. Diabetes Technol Ther. 2008 Oct;10(5):377-83. doi: 10.1089/dia.2008.0068. PMID 18715214
- [Background] Hermanides J, Norgaard K, Bruttomesso D, Mathieu C, Frid A, Dayan CM, Diem P, Fermon C, Wentholt IM, Hoekstra JB, DeVries JH. Sensor-augmented pump therapy lowers HbA(1c) in suboptimally controlled Type 1 diabetes; a randomized controlled trial. Diabet Med. 2011 Oct;28(10):1158-67. doi: 10.1111/j.1464-5491.2011.03256.x. PMID 21294770
- [Background] JDRF CGM Study Group. JDRF randomized clinical trial to assess the efficacy of real-time continuous glucose monitoring in the management of type 1 diabetes: research design and methods. Diabetes Technol Ther. 2008 Aug;10(4):310-21. doi: 10.1089/dia.2007.0302. PMID 18828243
- [Background] Rickels MR, Schutta MH, Mueller R, Markmann JF, Barker CF, Naji A, Teff KL. Islet cell hormonal responses to hypoglycemia after human islet transplantation for type 1 diabetes. Diabetes. 2005 Nov;54(11):3205-11. doi: 10.2337/diabetes.54.11.3205. PMID 16249446
- [Background] Rickels MR, Schutta MH, Mueller R, Kapoor S, Markmann JF, Naji A, Teff KL. Glycemic thresholds for activation of counterregulatory hormone and symptom responses in islet transplant recipients. J Clin Endocrinol Metab. 2007 Mar;92(3):873-9. doi: 10.1210/jc.2006-2426. Epub 2006 Dec 27. PMID 17192287
- [Derived] Rickels MR, Peleckis AJ, Dalton-Bakes C, Naji JR, Ran NA, Nguyen HL, O'Brien S, Chen S, Lee I, Schutta MH. Continuous Glucose Monitoring for Hypoglycemia Avoidance and Glucose Counterregulation in Long-Standing Type 1 Diabetes. J Clin Endocrinol Metab. 2018 Jan 1;103(1):105-114. doi: 10.1210/jc.2017-01516. PMID 29190340

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Intervention Group (Group 1) consists of participants with Type 1 Diabetes complicated by Hypoglycemia Unawareness.
  There were two Control Groups:
  (Group 2) T1Ds With Intact Awareness and (Group 3) Non-diabetics are used as a baseline for clinical significance. Neither of these two Control Groups wore a CGM nor were they analyzed at 6-month and 18-month time-points.
Groups:
- Hypoglycemia Unaware T1 Diabetics: This Intervention Group (Group 1) consists of participants with type 1 diabetes complicated by hypoglycemia unawareness. Patients wore an RT-CGM for 18 months. We studied glucose production and symptom generation during insulin-induced hypoglycemia (metabolic testing) by subjecting this intervention group to a pair of metabolic clamps (hypoglycemic and euglycemic) at baseline, at 6 months and at 18 months to determine if hypoglycemia avoidance can reverse unawareness.
- Control Group 2 - T1Ds With Intact Awareness; Control Group 3 - Non-diabetics: This control group was one of two control groups used as a baseline for clinical significance. Neither of these two control groups wore a CGM nor were they analyzed at 6-month and 18-month time-points.
Period: Overall Study
Arm/Group | Hypoglycemia Unaware T1 Diabetics | Control Group 2 - T1Ds With Intact Awareness | Control Group 3 - Non-diabetics
Started | 13 | 12 | 12
Completed | 11 | 11 | 12
Not Completed | 2 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Did not meet inclusion | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Hypoglycemia Unaware T1 Diabetics are the intervention group. The 2 control groups (Non-diabetics & T1Ds with intact Awareness) were used for clinical significance and were not assessed for outcome measures. These control group numbers have been included in the participant Flow, Baseline Characteristics and Adverse Events modules only.
Groups:
- Hypoglycemia Unaware T1 Diabetics: This main arm is the intervention group. It consists of participants with type 1 diabetes complicated by hypoglycemia unawareness. Patients wore an RT-CGM for 18 months. We studied glucose production and symptom generation during insulin-induced hypoglycemia (metabolic testing) by subjecting this intervention group to a pair of metabolic clamps (hypoglycemic and euglycemic) at baseline, at 6 months and at 18 months to determine if hypoglycemia avoidance can reverse unawareness.
  RT-CGM: Each device is approximately the size of a pager and transmits with a subcutaneously placed sensor consisting of a 21 - 26 gauge needle 5 - 12 mm in length. Sensors are placed using sterile precautions and changed every 3 - 7 days depending on the manufacturers' instructions. All devices are approved as adjunctive tools to blood glucose monitoring that will be continued at least 4 times daily, before each meal and at bedtime.
- Control Group 2 - T1Ds With Intact Awareness: Control Group 2 consists of 12 type one diabetics with intact awareness. Participants in control group 2 are enrolled as a baseline for clinical significance and not assessed for outcome measures. Control group 2 did not wear a CGM. They attended 3 visits (screening, HypoGlycemic clamp and EuGlycemic clamp) and they were not analyzed at 6-month and 18-month time-points.
- Control Group 3 - Non-diabetics: Control Group 3 consists of 12 non-diabetics. Participants in control group 3 are enrolled as a baseline for clinical significance and not assessed for outcome measures. Control group 3 did not wear a CGM. They attended 3 visits (screening, HypoGlycemic clamp and EuGlycemic clamp) and they were not analyzed at 6-month and 18-month time-points.
- Total: Total of all reporting groups
Arm/Group | Hypoglycemia Unaware T1 Diabetics | Control Group 2 - T1Ds With Intact Awareness | Control Group 3 - Non-diabetics | Total
Number analyzed (Participants) | 13 | 12 | 12 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 12 | 37
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Hypoglycemia Unaware T1 Diabetes RT-CGM
  years | 46.307 (14.343) | 35.416 (12.442) | 46.166 (7.309) | 42.729 (12.593)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 6 | 18
  Male | 5 | 8 | 6 | 19
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 12 | 37

OUTCOME MEASURES:

1. Primary Outcome: Endogenous Glucose Production
Description: Measure of hepatic glucose output during final hour of hypoglycemic clamp.
  Outcome Measures are not assigned to the control groups in ct.gov as they were only used as a baseline for clinical significance. Neither group wore a CGM nor were they analyzed at 6-month and 18-month time-points.
Time Frame: 6 months
Population: Type 1 Diabetes with Hypoglycemia Unawareness. Patients wear an RT-CGM for 18 months.
Measure: Mean (Standard Error); unit: mg/kg/min
Groups:
- Hypoglycemia Unaware T1 Diabetes RT-CGM: This arm is the intervention group. It consists of participants with type 1 diabetes complicated by hypoglycemia unawareness. Patients wore an RT-CGM for 18 months. We studied glucose production and symptom generation during insulin-induced hypoglycemia (metabolic testing) by subjecting this intervention group to a pair of metabolic clamps (hypoglycemic and euglycemic) at baseline, at 6 months and at 18 months to determine if hypoglycemia avoidance can reverse unawareness.
  Please note: Arms are not assigned to the two control groups (non-diabetics and T1Ds with intact awareness) in ct.gov as they are only used as a baseline for clinical significance. Neither group wore a CGM nor are they analyzed at 6-month and 18-month time-points.
  RT-CGM: Each device is approximately the size of a pager and transmits with a subcutaneously placed sensor consisting of a 21 - 26 gauge needle 5 - 12 mm in length. Sensors are placed using sterile precautions and changed every 3 - 7 days depending on the manufacturers' instructions. All devices are approved as adjunctive tools to blood glucose monitoring that will be continued at least 4 times daily, before each meal and at bedtime.
Arm/Group | Hypoglycemia Unaware T1 Diabetes RT-CGM
Number analyzed (Participants) | 13
mg/kg/min | 0.54 (0.07)

2. Secondary Outcome: Endogenous Glucose Production
Description: Measure of hepatic glucose output during final hour of hypoglycemic clamp
Time Frame: 18 months
Population: Type 1 Diabetes with Hypoglycemia Unawareness. Patients wear an RT-CGM for 18 months.
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Hypoglycemia Unaware T1 Diabetes RT-CGM
Number analyzed (Participants) | 11
mg/kg/min | 0.84 (0.15)

3. Secondary Outcome: Autonomic Symptom Response to Hypoglycemia
Description: Response measure during hypoglycemic clamp using an Autonomic Symptom Questionnaire.
  The autonomic symptom response is calculated during the final hour of the Hypoglycemic clamp as the sum of scores ranging from 0 (none) to 5 (severe) for each of the following symptoms: anxiety, palpitations, sweating, tremor, hunger, and tingling. This results in a minimum of 0 or a maximum of 30 score with the higher score a better outcome. The scale title is Autonomic Symptom Response to hypoglycemia.
Time Frame: 6 months
Population: Type 1 Diabetes with Hypoglycemia Unawareness. Patients wear an RT-CGM for 18 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hypoglycemia Unaware T1 Diabetes RT-CGM
Number analyzed (Participants) | 13
score on a scale | 5.1 (1.0)

4. Secondary Outcome: Autonomic Symptom Response to Hypoglycemia
Description: as for outcome 3
Time Frame: 18 months
Population: Type 1 Diabetes with Hypoglycemia Unawareness. Patients wear an RT-CGM for 18 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hypoglycemia Unaware T1 Diabetes RT-CGM
Number analyzed (Participants) | 11
score on a scale | 5.6 (1.2)

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse event and/or serious adverse event definitions do not differ from those of clinical trials.gov
Groups:
- Hypoglycemia Unaware T1 Diabetics: This main arm is the intervention group. It consists of participants with type 1 diabetes complicated by hypoglycemia unawareness. Patients wore an RT-CGM for 18 months. We studied glucose production and symptom generation during insulin-induced hypoglycemia (metabolic testing) by subjecting this intervention group to a pair of metabolic clamps (hypoglycemic and euglycemic) at baseline, at 6 months and at 18 months to determine if hypoglycemia avoidance can reverse unawareness.
  RT-CGM: Each device is approximately the size of a pager and transmits with a subcutaneously placed sensor consisting of a 21 to 26-gauge needle 5 to12 mm in length. Sensors are placed using sterile precautions and changed every 3 to 7 days depending on the manufacturers' instructions. All devices are approved as adjunctive tools to blood glucose monitoring that will be continued at least 4 times daily, before each meal and at bedtime.
- Control Group 2 - T1 Diabetics: Control Group 2 consists of 12 type one diabetics with intact awareness. Participants in control group 2 are enrolled as a baseline for clinical significance and not assessed for outcome measures. Control group 2 did not wear a CGM. They attended 3 visits (screening, HypoGlycemic clamp and EuGlycemic clamp) and they were not analyzed at 6-month and 18-month time-points.
- Control Group 3 - Non Diabetics: Control Group 3 consists of 12 non-diabetics. Participants in control group 3 are enrolled as a baseline for clinical significance and not assessed for outcome measures. Control group 3 did not wear a CGM. They attended 3 visits (screening, HypoGlycemic clamp and EuGlycemic clamp) and they were not analyzed at 6-month and 18-month time-points.
Arm/Group | Hypoglycemia Unaware T1 Diabetics | Control Group 2 - T1 Diabetics | Control Group 3 - Non Diabetics
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No